CLINICAL TRIAL: NCT06046144
Title: Comparison of 3 in Vivo Microscopic Imaging Techniques for the Diagnosis of Pigmented Tumors. Monocentric Retrospective Study of 170 Tumors
Brief Title: Comparison of 3 in Vivo Microscopic Imaging Techniques for the Diagnosis of Pigmented Tumors
Acronym: Micro3
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1142023/CHUSTE
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-08

CONDITIONS: Basal Cell Carcinoma; Lentigo Maligna; Melanoma; Nevus; Seborrheic Keratosis; Lentigo
Keywords: Melanoma diagnosis; Diagnosis Imaging; Fluorescence-Advanced videodermatoscopy; Reflectance confocal microscopy; Super-high magnification dermoscopy
MeSH Terms: conditions — Carcinoma, Basal Cell; Hutchinson's Melanotic Freckle; Melanoma; Nevus; Keratosis, Seborrheic; Lentigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a pigmented skin lesion: Patients with a pigmented skin lesion of more than 3mm diameter which have benefited systematically of all 3 imaging techniques at the same time, followed by either a surgical excision or annual imaging monitoring.
  Interventions: Diagnostic Test: Fluorescence-Advanced videodermatoscopy; Diagnostic Test: Reflectance confocal microscopy; Diagnostic Test: Super-high magnification dermoscopy

INTERVENTIONS:
Diagnostic Test: Fluorescence-Advanced videodermatoscopy — Datas collected : Presence or absence of atypical roundish cell, dendritic cell, atypical nests, points, folliculotropism, blue homogenous zone, regular honeycomb pattern.
  Between 10 and 60 images taken by a hand-held camera set directly on the skin lesion, with an oily interface.
Diagnostic Test: Reflectance confocal microscopy — Datas collected : Presence or absence of atypical roundish cell, dendritic cell, atypical nests, points, folliculotropism, blue homogenous zone, regular honeycomb pattern.
  Between 10 and 60 images taken by a hand-held camera set directly on the skin lesion, with an oily interface.
Diagnostic Test: Super-high magnification dermoscopy — Datas collected : Presence or absence of atypical roundish cell, dendritic cell, atypical nests, points, folliculotropism, blue homogenous zone, regular honeycomb pattern.
  Between 10 and 60 images taken by a hand-held camera set directly on the skin lesion, with an oily interface.

SUMMARY:
Reflectance confocal microscopy (RCM) is the reference in vivo imaging technique for identifying malignant melanocytic tumors prior to surgical excision. However, it is not widely used due to its high cost and highly technical and time-consuming nature.

In addition to Reflectance confocal microscopy (RCM), it currently use 2 less expensive dermatoscopes that also allow in vivo diagnosis: super-high magnification dermoscopy (D400) and Fluorescence-Advanced videodermatoscopy (FAV).

DETAILED DESCRIPTION:
Several studies have demonstrated their interest in the in vivo diagnosis of melanocytic tumors, but without any comparison between these methods.

In our current practice, many patients have benefited from these 3 imaging modalities for benign and malignant lesions.

Therefore, our aim is to analyze these images and compare their performance in the diagnosis of benign and malignant pigmented lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pigmented skin lesion of more than 3mm diameter which have benefited systematically of all 3 imaging techniques at the same time, followed by either a surgical excision or annual imaging monitoring.

Exclusion Criteria:

* Bad quality images
* Insufficient number of images
* Uncertain diagnosis given by the pathologist
* Refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a pigmented skin lesion of more than 3mm diameter which have benefited systematically of all 3 imaging techniques at the same time, followed by either a surgical excision or annual imaging monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
To compare the the relevance of each technique for the diagnostic of pigmented lesions. | Day 1
  The nature of the tumor is diagnosed by the imaging technique.

SECONDARY OUTCOMES:
Comparison of performance of imaging techniques | Day 1
  Analyze the results of imaging of each technique.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc PERROT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No